CLINICAL TRIAL: NCT02871635
Title: BI 695501 Versus Humira® in Patients With Active Crohn's Disease: a Randomized, Double-blind, Multicenter, Parallel Group, Exploratory Trial Comparing Efficacy, Endoscopic Improvement, Safety, and Immunogenicity
Brief Title: BI 695501 Versus Humira in Patients With Active Crohn's Disease: a Trial Comparing Efficacy, Endoscopic Improvement, Safety, and Immunogenicity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1297.4; 2016-000612-14 (EudraCT Number)
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — BI 695501; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BI 695501 (Experimental)
  Interventions: Drug: BI 695501
- HUMIRA + BI 695501 (Active Comparator)
  Interventions: Drug: BI 695501; Drug: HUMIRA

INTERVENTIONS:
Drug: BI 695501
Drug: HUMIRA
  Arms: HUMIRA + BI 695501

SUMMARY:
Primary Objective:

The primary objective of this trial is to compare the clinical efficacy of BI 695501 with EU-approved Humira® in patients with active Crohn's disease (CD).

Secondary Objectives:

The secondary objectives of this trial are to compare the efficacy and safety of BI 695501 with EU-approved Humira® across the induction and maintenance phases.

ELIGIBILITY:
Inclusion criteria:

* Males and females aged >=18 and =<80 years at Screening who have a diagnosis of moderate to severely active Crohn's Disease (CD), confirmed by endoscopy or radiologic evaluation, for more than 4 months with evidence of mucosal ulceration. Patients must have all of the following:

  * Crohn's Disease Activity Index (CDAI) score of >=220 and =<450
  * A diagnosis of Crohn's Disease (CD) confirmed by ileocolonoscopy during Screening
  * Presence of mucosal ulcers in at least one segment of the ileum or colon and a SES-CD score ≥7 (for patients with isolated ileal disease SES-CD score ≥4), as assessed by ileocolonoscopy and confirmed by central independent reviewer(s) before randomization
* Anti-tumor necrosis factor (TNF) patients or patients previously treated with infliximab who had initially responded and who meet one of the following criteria:

  * Responded and developed secondary resistance due confirmed anti-infliximab anti-drug antibody formation, which caused infliximab depletion
  * Responded and became intolerant
* Further inclusion criteria apply

Exclusion criteria:

* Patients with ulcerative colitis or indeterminate colitis
* Patients with symptomatic known obstructive strictures
* Surgical bowel resection performed within 6 months prior to Screening or planned resection at any time while enrolled in the trial
* Patients with an ostomy or ileoanal pouch
* Patients with short bowel syndrome
* Patients who have previously used infliximab and have never clinically responded
* Patients who have previously received treatment with adalimumab, or who have participated in an adalimumab or adalimumab biosimilar clinical trial
* Further exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (92):
- United States (19):
  - Borland-Groover Clinic, Jacksonville, Florida
  - Hope Clinical Research, Kissimmee, Florida
  - Center for Advanced GI, Maitland, Florida
  - Advance Medical Research Center, Miami, Florida
  - Advanced Research Institute, Inc, New Port Richey, Florida
  - Doctors Clinical Research, East Point, Georgia
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - MGG Group Co. Inc. / Chevy Chase Clinical Research,, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Healthcare Research Network, Hazelwood, Missouri
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Houston Endoscopy and Research Center, Houston, Texas
  - Biopharma Informatic, Inc, dba Research Consultants, Katy, Texas
  - Sagact, Pllc, San Antonio, Texas
  - Baylor Scott and White Healthcare, Temple, Texas
  - Victoria Gastroenterology, Victoria, Texas
- Belarus (3):
  - Gomel Regional Clinical, Homyel
  - City Clinical Hospital # 10, Minsk
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- University Clinical Centre Sarajevo, Sarajevo, Bosnia and Herzegovina
- Croatia (2):
  - Clinical Hospital Osijek, Osijek
  - Polyclinic Bonifarm, Zagreb
- Czechia (12):
  - Vojenska nemocnice Brno, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - CTCenter Mave, s.r.o., Cllinical Trials Center, Olomouc, Olomouc
  - Gregar s.r.o., Olomouc
  - PreventaMed, s.r.o., Olomouc
  - University Hospital Ostrava, Ostrava-Poruba
  - Vitkovice Hospital, Ostrava-Vitkovice
  - Medicon, a.s., Prague
  - Axon Clinical, s.r.o., Prague
  - University Hospital Na Bulovce, Prague
  - General Hospital Pribram, Příbram
  - Masaryk Hospital, Internal Department, Ústí nad Labem
- Crohn Colitis Centrum Rhein Main, Frankfurt, Germany
- Greece (3):
  - General Hospital of Athens Evangelismos, Athens
  - University General Hospital of Heraklion, Heraklion, Crete
  - General Hospital of Rhodes, Rhodes
- Israel (6):
  - Haemek Medical Center, Afula
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center Tel Hashomer, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Poland (11):
  - KLIMED Marek Klimkiewicz, Bialystok
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Polimedica Centrum Badan, Kielce
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Medical Center Pleiades, Krakow
  - SANTA FAMILIA Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Clinic Medical Center; Nowa Sol, Nowa Sól
  - Ai Medical Center, private practice, Poznan, Poznan
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Specialized Medical Practice. Dr med. Marek Horynski, Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
- Russia (14):
  - Multidisciplinary Medical Clinic "Anthurium", Barnaul
  - GUZ Reg. Clinical Hospital, Kemerovo, Kemerovo
  - Clinical Hospital No. 24, Moscow, Moscow
  - Murmansk Regional Clinical Hospital named after Bayandin, Murmansk
  - Reg.Clin.Hosp.n.a.Semashko, Nizhny Novgorod
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - FSBSI "Scientific and Research Institute of Physiology and Basic Medicine", Novosibirsk
  - BHI of Omsk region - Clinical Oncology Dispensary, Omsk
  - SBIH City Clinical Hospital #31, Saint Petersburg
  - Baltic Med,LLC Clinic BaltMed Ozerki, Saint Petersburg
  - EKO-Bezopasnost, St. Petersburg, Saint Petersburg
  - LLC IClinic, Saint Petersburg
  - Private Educational Institution of Higher Education "Medical University "REAVIZ", Samara
  - NonState Healthcare Institution Central Clinical Hospital, Samara station JSC "Russian Railways", Samara
- Serbia (5):
  - Clinical Medical Center Zvezdara, Belgrade, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska kosa, Belgrade, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty, Ankara
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital, Gaziantep
  - Kartal Lutfi Kirdar Research and Training Hospital, Istanbul
  - Kocaeli University Research and Training Hospital, Kocaeli
- Ukraine (9):
  - CI Cherkasy RH of Cherkasy Reg.Council, Cherkasy
  - CHI Prof.O.O.Shalimov Kharkiv City Clinical Hospital #2, Kharkiv
  - Med Center 'Ok!Clinic+' of International Institute of Clinical Trials LLC, Kiev
  - Private Enterprise Private Manufacturing Company "Acinus", Kirovohrad
  - Medical Center Medical Clinic Kyiv, Kyiv
  - Clin Hosp.8 P.L.Shupyk NMA of PGE, Kyiv
  - Vinnytsia M.I. Pyrogov NMU Ch of internal medicine #3, Vinnytsia
  - M.I. Pyrogov VRCH, Vinnytsia, Vinnytsia
  - Clin.Hosp#1,Zaporizhzhia, Zaporizhzhia
- United Kingdom (2):
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Walsall Manor Hospital, Walsall

REFERENCES:
- [Derived] Strand V. Summary of Research: Immunogenicity of Adalimumab Reference Product and Adalimumab-adbm in Patients with Rheumatoid Arthritis, Crohn's Disease, and Chronic Plaque Psoriasis: A Pooled Analysis of the VOLTAIRE trials. Rheumatol Ther. 2025 Aug;12(4):613-616. doi: 10.1007/s40744-025-00766-6. Epub 2025 Jun 11. PMID 40498294
- [Derived] Strand V, McCabe D, Bender S. Immunogenicity of adalimumab reference product and adalimumab-adbm in patients with rheumatoid arthritis, Crohn's disease and chronic plaque psoriasis: a pooled analysis of the VOLTAIRE trials. BMJ Open. 2024 Nov 17;14(11):e081687. doi: 10.1136/bmjopen-2023-081687. PMID 39551590
- [Derived] Hanauer S. Plain language summary of the VOLTAIRE-CD study in people with moderate-to-severe active Crohn's disease. Immunotherapy. 2022 Dec;14(17):1353-1359. doi: 10.2217/imt-2022-0129. Epub 2022 Dec 13. PMID 36511191
- [Derived] Hanauer S, Liedert B, Balser S, Brockstedt E, Moschetti V, Schreiber S. Safety and efficacy of BI 695501 versus adalimumab reference product in patients with advanced Crohn's disease (VOLTAIRE-CD): a multicentre, randomised, double-blind, phase 3 trial. Lancet Gastroenterol Hepatol. 2021 Oct;6(10):816-825. doi: 10.1016/S2468-1253(21)00252-1. Epub 2021 Aug 11. PMID 34388360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an exploratory, randomized, 56-week, double-blind, parallel arm, multiple dose, active comparator trial of BI 695501 and EU-approved Humira, with a 48-week treatment period and a 10-week follow-up period (starting after last dose of trial medication at Week 46) in patients with moderately to severely active Crohn's Disease (CD)
Pre-assignment Details: The trial consisted of a screening period of up to a maximum of 28 days, a 48-week treatment period consisting of an induction period from baseline to Week 4 and a maintenance period from Week 5 to Week 48, and a 10-week safety follow-up period (starting after last dose of trial medication at Week 46).
Groups:
- BI 695501: Patients randomized to BI 695501 received treatment every 2 weeks until Week 4 when they were assessed for clinical response. If classified as responders (Crohn's Disease Activity Index (CDAI) decrease of ≥70 compared to baseline), patients continued to receive BI 695501 every 2 weeks until the end of the treatment (EoT) period (Week 46).
  Patients were administered with a loading dose of 160 milligram (mg) BI 695501 on Day 1, followed by 80 mg BI 695501 2 weeks later (Day 15), and thereafter 40 mg BI 695501 every 2 weeks until Week 46. Trial medication was administered by subcutaneous (SC) injection.
- Humira EU: Patients randomized to EU-approved Humira received treatment every 2 weeks until Week 4 when they were assessed for clinical response. If classified as responders, patients continued to receive EU-approved Humira until Week 22 and then switched to receive BI 695501 every 2 weeks from Week 24 until the EoT period (Week 46).
  Patients were administered with a loading dose of 160 mg EU-approved Humira on Day 1, followed by 80 mg EU-approved Humira 2 weeks later (Day 15), and 40 mg EU-approved Humira every 2 weeks until Week 22. Patients were then switched to receive 40 mg BI 695501 every 2 weeks from Week 24 until Week 46. Trial medication was administered by SC injection.
Period: Overall Study
Arm/Group | BI 695501 | Humira EU
Started | 72 | 75
Completed | 54 | 56
Not Completed | 18 | 19
Not completed — Primary lack of efficacy | 4 | 4
Not completed — Protocol Violation | 3 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Pregnancy | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 4 | 4
Not completed — Secondary lack of efficacy | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAF) contained all randomized patients who received at least 1 dose (full or partial) of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695501 | Humira EU | Total
Number analyzed (Participants) | 72 | 75 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (13.44) | 33.2 (11.52) | 35.3 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 39 | 44 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 69 | 67 | 136
  Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 69 | 74 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Crohn's Disease Activity Index score at baseline [Mean (Standard Deviation); unit: Scores on a scale] — Crohn's Disease Activity Index (CDAI) is a valid instrument to measure severity in Crohn's disease. The CDAI is composed of 8 factors (Number of liquid stools, abdominal pain, general well being, extra-intestinal complications, antidiarrheal drugs, abdominal mass, hematocrit, body weight) the score is calculated by adding up the scores after adjustment with a weighting factor. The total score ranges from 0 to approx. 600, higher scores indicates more severe disease. A score of less than or equal to 150 is evaluated as a remission while 220 and 450 indicate moderate to severely active disease.
  Scores on a scale | 307.3 (76.69) | 303.6 (64.39) | 305.4 (70.46)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Clinical Response (CDAI Decrease of ≥70 Compared With Baseline) at Week 4
Description: The Crohn's Disease Activity Index (CDAI) is a validated instrument to measure disease severity in Crohn's Disease (CD). The CDAI score is a sum of the 8 factors (number of liquid stools, abdominal pain, general well-being, extra-intestinal complications, antidiarrheal drugs, abdominal mass, hematocrit and body weight) after adjustment with a weighting factor. Higher CDAI scores indicating more active disease.
  The CDAI decrease at Week 4 was assessed as the decrease relative to baseline measurement, patients with a decrease ≥70 were responders.
  Percentage=least squares means per treatment group back transformed using inverse logit function. Missing data were imputed according to non-responder imputation (NRI) and last observation carried forward (LOCF).
Time Frame: Week 4
Population: The full analysis set (FAS) contained all randomized patients who received at least 1 dose of trial medication, and had all efficacy measures relevant for the CDAI, measured at baseline and at least once postbaseline.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 68 | 72
Percentage of participants | 88.0 | 93.1
Statistical Analysis 1: Comparison: BI 695501 vs Humira EU; Was analyzed using a log-linked binomial model, described as: response to treatment at Week 4 = treatment+prior infliximab exposure+screening Simple Endoscopic Score for Crohn's Disease (SES-CD); Test type: Other; Risk Ratio (RR) = 0.945, 90% CI 2-sided [0.870 to 1.028] — BI 695501 as numerator Humira EU as denominator
Statistical Analysis 2: Comparison: BI 695501 vs Humira EU; Was to be analyzed using a log-linked binomial model, described as: response to treatment at Week 4 = treatment+prior infliximab exposure+screening Simple Endoscopic Score for Crohn's Disease (SES-CD); Test type: Other; Risk Ratio (RR) = 0.945, 95% CI 2-sided [0.856 to 1.044] — BI 695501 as numerator Humira EU as denominator

2. Secondary Outcome: Percentage of Patients With a Clinical Response (CDAI Decrease of ≥70 Compared With Baseline) at Week 24
Description: The CDAI is a validated instrument to measure disease severity in CD. The CDAI score is a sum of the 8 factors (number of liquid stools, abdominal pain, general well-being, extra-intestinal complications, antidiarrheal drugs, abdominal mass, hematocrit and body weight) after adjustment with a weighting factor. Higher CDAI scores indicating more active disease.
  The CDAI decrease at Week 24 was assessed as the decrease relative to baseline measurement, patients with a decrease ≥70 were responders.
  Percentage=least squares means per treatment group back transformed using inverse logit function. Missing data were imputed according to NRI and LOCF.
Time Frame: Week 24
Population: The FAS contained all randomized patients who received at least 1 dose of trial medication, and had all efficacy measures relevant for the CDAI, measured at baseline and at least once postbaseline.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 68 | 72
Percentage of participants | 87.4 | 87.4
Statistical Analysis 1: Comparison: BI 695501 vs Humira EU; Was to be analyzed using a log-linked binomial model, described as: response to treatment at Week 24 = treatment+prior infliximab exposure+screening Simple Endoscopic Score for Crohn's Disease (SES-CD); Test type: Other; Risk Ratio (RR) = 1.000, 90% CI 2-sided [0.871 to 1.148] — BI 695501 as numerator Humira EU as denominator
Statistical Analysis 2: Comparison: BI 695501 vs Humira EU; [analysis description as in outcome 2, analysis 1]; Test type: Other; Risk Ratio (RR) = 1.000, 95% CI 2-sided [0.848 to 1.178] — BI 695501 as numerator Humira EU as denominator

3. Secondary Outcome: Percentage of Patients in Clinical Remission (CDAI <150) at Week 24
Description: The CDAI is a validated instrument to measure disease severity in CD. The CDAI score is a sum of the 8 factors (number of liquid stools, abdominal pain, general well-being, extra-intestinal complications, antidiarrheal drugs, abdominal mass, hematocrit and body weight) after adjustment with a weighting factor. Higher CDAI scores indicating more active disease.
  Patients with CDAI <150 at Week 24 were considered as clinical remission cases. Percentage=least squares means per treatment group back transformed using inverse logit function. Missing data were imputed according to NRI and LOCF.
Time Frame: at Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 68 | 72
Percentage of participants | 68.6 | 76.2
Statistical Analysis 1: Comparison: BI 695501 vs Humira EU; [analysis description as in outcome 2, analysis 1]; Test type: Other; Risk Ratio (RR) = 0.900, 90% CI 2-sided [0.751 to 1.078] — BI 695501 as numerator Humira EU as denominator
Statistical Analysis 2: Comparison: BI 695501 vs Humira EU; [analysis description as in outcome 2, analysis 1]; Test type: Other; Risk Ratio (RR) = 0.9000, 95% CI 2-sided [0.725 to 1.116] — BI 695501 as numerator Humira EU as denominator

4. Secondary Outcome: Percentage of Patients With Adverse Events (AEs), Serious AEs (SAEs), and AEs of Special Interest (AESIs)
Description: Analysis of AEs focused on treatment-emergent AEs (TEAEs). For the period 1 'Baseline - Week 24', TEAEs were defined as AEs that started or worsened on or after first dose of trial medication and prior to date of the Week 24 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients who discontinued treatment before Week 24. For the period 2 'Week 24 - Week 46', TEAEs were defined as AEs that started or worsened on Week 24 visit and prior to or on Week 56 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients discontinuing treatment prior to Week 46. TEAEs and SAEs (including investigator-assessed trial medication-related TEAEs) and AESIs are reported. The following were considered an AESI: hepatic injury, anaphylactic reactions, serious infection and hypersensitivity reactions.
Time Frame: From first administration of trial medication until 10 weeks after last administration, up to a maximum of 56 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 72 | 75
Percentage of participants
  TEAE -Period 1 | 62.5 | 56.0
  serious TEAE - Period 1 | 8.3 | 10.7
  AESI TEAE - Period 1 | 2.8 | 2.7
  TEAE - Period 2 | 43.1 | 45.3
  serious TEAE - Period 2 | 2.8 | 12.0
  AESI TEAE - Period 2 | 2.8 | 2.7

5. Secondary Outcome: Percentage of Patients With Infections
Description: The percentage of patients with TEAEs for infections are reported. For the period 1 'Baseline - Week 24', TEAEs were defined as AEs that started or worsened on or after first dose of trial medication and prior to date of the Week 24 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients who discontinued treatment before Week 24. For the period 2 'Week 24 - Week 46', TEAEs were defined as AEs that started or worsened on Week 24 visit and prior to or on Week 56 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients discontinuing treatment prior to Week 46.
Time Frame: From first administration of trial medication until 10 weeks after last administration, up to a maximum of 56 weeks.
Population: The SAF contained all randomized patients who received at least 1 dose (full or partial) of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 72 | 75
Percentage of participants
  Period 1 | 23.6 | 22.7
  Period 2 | 19.4 | 22.7

6. Secondary Outcome: Percentage of Patients With Serious Infections
Description: The percentage of patients with TEAEs for serious infections are reported. For the period 1 'Baseline - Week 24', TEAEs were defined as AEs that started or worsened on or after first dose of trial medication and prior to date of the Week 24 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients who discontinued treatment before Week 24. For the period 2 'Week 24 - Week 46', TEAEs were defined as AEs that started or worsened on Week 24 visit and prior to or on Week 56 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients discontinuing treatment prior to Week 46.
Time Frame: From first administration of trial medication until 10 weeks after last administration, up to a maximum of 56 weeks.
Population: The SAF contained all randomized patients who received at least 1 dose (full or partial) of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 72 | 75
Percentage of participants
  Period 1 | 2.8 | 2.7
  Period 2 | 1.4 | 4.0

7. Secondary Outcome: Percentage of Patients Who Experienced Hypersensitivity Reactions
Description: The percentage of patients with TEAEs for hypersensitivity reactions is reported. For the period 1 'Baseline - Week 24', TEAEs were defined as AEs that started or worsened on or after first dose of trial medication and prior to date of the Week 24 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients who discontinued treatment before Week 24. For the period 2 'Week 24 - Week 46', TEAEs were defined as AEs that started or worsened on Week 24 visit and prior to or on Week 56 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients discontinuing treatment prior to Week 46.
Time Frame: From first administration of trial medication until 10 weeks after last administration, up to a maximum of 56 weeks.
Population: The SAF contained all randomized patients who received at least 1 dose (full or partial) of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 72 | 75
Percentage of participants
  Period 1 | 5.6 | 2.7
  Period 2 | 2.8 | 6.7

8. Secondary Outcome: Percentage of Patients Who Experienced Drug Induced Liver Injury (DILI)
Description: The percentage of patients with TEAEs for DILIs is reported. For the period 1 'Baseline - Week 24', TEAEs were defined as AEs that started or worsened on or after first dose of trial medication and prior to date of the Week 24 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients who discontinued treatment before Week 24. For the period 2 'Week 24 - Week 46', TEAEs were defined as AEs that started or worsened on Week 24 visit and prior to or on Week 56 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients discontinuing treatment prior to Week 46.
Time Frame: From first administration of trial medication until 10 weeks after last administration, up to a maximum of 56 weeks.
Population: The SAF contained all randomized patients who received at least 1 dose (full or partial) of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 72 | 75
Percentage of participants
  Period 1 | 0.0 | 0.0
  Period 2 | 0.0 | 0.0

9. Secondary Outcome: Percentage of Patients With Injection Site Reactions
Description: The percentage of patients with TEAEs for injection site reactions is reported. For the period 1 'Baseline - Week 24', TEAEs were defined as AEs that started or worsened on or after first dose of trial medication and prior to date of the Week 24 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients who discontinued treatment before Week 24. For the period 2 'Week 24 - Week 46', TEAEs were defined as AEs that started or worsened on Week 24 visit and prior to or on Week 56 visit or within 10 weeks (70 days, inclusive) after last dose of trial medication for patients discontinuing treatment prior to Week 46.
Time Frame: From first administration of trial medication until 10 weeks after last administration, up to a maximum of 56 weeks.
Population: The SAF contained all randomized patients who received at least 1 dose (full or partial) of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501 | Humira EU
Number analyzed (Participants) | 72 | 75
Percentage of participants
  Period 1 | 0.0 | 6.7
  Period 2 | 1.4 | 1.3

ADVERSE EVENTS:
Time Frame: From first administration of trial medication until 10 weeks after last administration, up to a maximum of 56 weeks.
Description: The Safety Analysis Set (SAF) contained all randomized patients who received at least 1 dose (full or partial) of trial medication.
Groups:
- BI 695501 (Baseline - Week 24 + 10 Weeks [70 Days]); BI 695501 (Week 24 - Week 46 + 10 Weeks [70 Days]): Patients randomized to BI 695501 received treatment every 2 weeks until Week 4 when they were assessed for clinical response. If classified as responders (CDAI decrease of ≥70 compared to baseline), patients continued to receive BI 695501 every 2 weeks until the end of the treatment (EoT) period (Week 46).
  Patients were administered with a loading dose of 160 milligram (mg) BI 695501 on Day 1, followed by 80 mg BI 695501 2 weeks later (Day 15), and thereafter 40 mg BI 695501 every 2 weeks until Week 46. Trial medication was administered by subcutaneous (SC) injection.
- Humira (Baseline - Week 24 + 10 Weeks [70 Days]); Humira (Week 24 - Week 46 + 10 Weeks [70 Days]): Patients randomized to EU-approved Humira received treatment every 2 weeks until Week 4 when they were assessed for clinical response. If classified as responders, patients continued to receive EU-approved Humira until Week 22 and then switched to receive BI 695501 every 2 weeks from Week 24 until the EoT period (Week 46).
  Patients were administered with a loading dose of 160 mg EU-approved Humira on Day 1, followed by 80 mg EU-approved Humira 2 weeks later (Day 15), and 40 mg EU-approved Humira every 2 weeks until Week 22. Patients were then switched to receive 40 mg BI 695501 every 2 weeks from Week 24 until Week 46. Trial medication was administered by SC injection.
Arm/Group | BI 695501 (Baseline - Week 24 + 10 Weeks [70 Days]) | Humira (Baseline - Week 24 + 10 Weeks [70 Days]) | BI 695501 (Week 24 - Week 46 + 10 Weeks [70 Days]) | Humira (Week 24 - Week 46 + 10 Weeks [70 Days])
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/75 | 0/72 | 0/75
Serious Adverse Events (participants affected / at risk) | 6/72 | 8/75 | 2/72 | 9/75
Other Adverse Events (participants affected / at risk) | 23/72 | 16/75 | 13/72 | 12/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (Baseline - Week 24 + 10 Weeks [70 Days]) (N=72) | Humira (Baseline - Week 24 + 10 Weeks [70 Days]) (N=75) | BI 695501 (Week 24 - Week 46 + 10 Weeks [70 Days]) (N=72) | Humira (Week 24 - Week 46 + 10 Weeks [70 Days]) (N=75)
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 2 | 5 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (Baseline - Week 24 + 10 Weeks [70 Days]) (N=72) | Humira (Baseline - Week 24 + 10 Weeks [70 Days]) (N=75) | BI 695501 (Week 24 - Week 46 + 10 Weeks [70 Days]) (N=72) | Humira (Week 24 - Week 46 + 10 Weeks [70 Days]) (N=75)
Respiratory tract infection (Infections and infestations) | 5 | 3 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 5 | 3
Crohn's disease (Gastrointestinal disorders) | 4 | 3 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 2 | 0
Weight increased (Investigations) | 4 | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT02871635/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT02871635/SAP_001.pdf